CLINICAL TRIAL: NCT00489671
Title: Differential Diagnosis Between Pancreatic Cancer and Chronic Pancreatitis: Value of the Detection of Urinary Cadmium
Brief Title: Urine Cadmium Levels in Predicting Pancreatic Cancer Risk in Patients With Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000550074; CCCWFU-98503; CCCWFU-BG03-223
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2015-10

CONDITIONS: Pancreatic Cancer; Precancerous Condition
Keywords: pancreatic cancer; precancerous condition
MeSH Terms: conditions — Pancreatic Neoplasms; Precancerous Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pre cancerous condition (pancreatitis)

SUMMARY:
RATIONALE: Measuring cadmium levels in urine samples from patients with chronic pancreatitis may help doctors predict which patients may develop pancreatic cancer. It may also help the study of cancer in the future.

PURPOSE: This clinical trial is studying urine cadmium levels in predicting pancreatic cancer risk in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Obtain urine samples and questionnaire data on cadmium exposure in patients with chronic pancreatitis.
* Analyze these data to determine risk of pancreatic cancer using urine cadmium levels.

Secondary

* Analyze these data in conjunction with data on serum CA 19-9, to determine whether urinary cadmium has clinical utility in predicting pancreatic cancer.
* Determine the sensitivity, specificity, and positive and negative predictive values for the cadmium test alone, CA 19-9 alone, and both tests together.

OUTLINE: This is a pilot study.

Patients complete a questionnaire over approximately 20 minutes on lifetime exposure to cadmium, including dietary, occupational, and recreational exposure, smoking history, and residence. Patients also provide a urine sample that is analyzed by atomic absorption spectrophotometry. Serum CA 19-9 levels are obtained from medical record if available.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical diagnosis of chronic pancreatitis
* Being seen in the Department of Gastroenterology at Wake Forest University Baptist Medical Center

PATIENT CHARACTERISTICS:

* No type II diabetes
* Able to understand and respond to questionnaire
* Able to provide urine specimen
* Speaks English

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chronic pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Exposure to cadmium, as measured by questionnaire data on dietary, occupational, and recreational exposure to cadmium, and by measurements of cadmium in urine | day 1
Risk of pancreatic cancer as determined by urine cadmium levels | day 1

SECONDARY OUTCOMES:
Predictive value of urinary cadmium on development of pancreatic cancer | day 1
Predictive value of urinary cadmium alone, CA 19-9 alone, and both tests together on development of pancreatic cancer | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gary G. Schwartz, MD, PhD, MPH, Study Chair — Wake Forest University Health Sciences